CLINICAL TRIAL: NCT03408444
Title: Evaluating Soft Contact Lens Prototypes for Myopia Control
Status: Completed | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5959
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (4):
- EMO-114 (Experimental): Test Lens 1
  Interventions: Device: EMO-114
- EMO-116 (Experimental): Test Lens 2
  Interventions: Device: EMO-116
- EMO-118 (Experimental): Test Lens 3
  Interventions: Device: EMO-118
- EMO-117 (Active Comparator): Test Lens 4
  Interventions: Device: EMO-117

INTERVENTIONS:
Device: EMO-114 — Subjects between the ages of 7 and 12 years old will be bilaterally fitted with one of the four types of test articles and wear lenses of the assigned lens type during the entire course of the study.
  Other Names: Test Lens 1
  Arms: EMO-114
Device: EMO-116 — Subjects between the ages of 7 and 12 years old will be bilaterally fitted with one of the four types of test articles and wear lenses of the assigned lens type during the entire course of the study.
  Other Names: Test Lens 2
  Arms: EMO-116
Device: EMO-118 — Subjects between the ages of 7 and 12 years old will be bilaterally fitted with one of the four types of test articles and wear lenses of the assigned lens type during the entire course of the study.
  Other Names: Test Lens 3
  Arms: EMO-118
Device: EMO-117 — Subjects between the ages of 7 and 12 years old will be bilaterally fitted with one of the four types of test articles and wear lenses of the assigned lens type during the entire course of the study.
  Other Names: Test Lens 4
  Arms: EMO-117

SUMMARY:
This is a multi-site, prospective, randomized, controlled, double-masked, four-arm-parallel-group, dispensing study. Each subject will be bilaterally fitted with one of four types of test articles and wear contact lenses of the assigned lens type during the entire course of the study. Test articles will be worn a minimum 8 hours per day and 5 days per week (subjects will be encouraged to wear study contact lenses 10 hours or more per day and 7 days per week) in a daily disposable modality for a minimum of 6 months and up to 1 year for a total of 7 scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read (or be read to), understand, and sign the Statement of Information and Assent and receive a fully executed copy of the form.
  2. The subject's parent(s) or legal guardian(s) must read, understand and sign the Statement of Informed Consent and receive a fully executed copy of the form.
  3. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  4. Between 7 and 12 years of age (inclusive).
  5. Have normal eyes (i.e., no ocular medications or infections of any type).
  6. Distance subjective best-sphere refraction must be between -0.75D and -4.50D (inclusive) in each eye.
  7. Cylindrical refraction must be 1.00D or less in each eye, by subjective sphero-cylindrical refraction.
  8. Have sphero-cylindrical best-corrected visual acuity of 20/25 (ie, 0.8 in decimal convention or 0.10 logMAR) or better in each eye.
  9. Cycloplegic objective sphero-cylindrical refraction (by auto refraction) must be between -0.75D and -4.50D in sphere and is 1.00D or less in cylinder in each eye (based on the average of 5 repeated sphero-cylindrical refraction measures).
  10. The difference in spherical equivalent power between the two eyes must be less than 1.50D (based on the average of 5 repeated sphero-cylindrical refraction measures).

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any systemic allergies, infectious disease (e.g., hepatitis, tuberculosis), autoimmune disease (e.g., rheumatoid arthritis), or other systemic diseases (e.g., diabetes), by the parent or legal guardian's report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear.
  4. Any current use of ocular topical medication.
  5. Any previous or planned ocular or intraocular surgery, including refractive surgery.
  6. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  7. Participation in any prior myopia control clinical study in the test group.
  8. Current or recent (within 30 days from enrollment) rigid lens wearers.
  9. History of orthokeratology treatment or use of other ophthalmic devices (e.g., bifocal, multifocal contact or spectacle lenses) or drugs (e.g., atropine or pirenzepine) for the purpose of controlling myopia progression.
  10. Any known hypersensitivity or allergic reaction to EyeCept® (or sponsor approved equivalent) Rewetting Drop Solution.
  11. Relatives of employee of investigational clinic (e.g., Investigator, Coordinator, Technician).
  12. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to, aphakia, uveitis, ocular hypertension, glaucoma, severe keratoconjunctivitis sicca, history of recurrent corneal erosions, keratoconus, keratoconus suspect, pellucid marginal degeneration, entropion, ectropion, extrusions, chalazia, and recurrent styes.
  13. Grade 3 or greater palpebral conjunctival observations or any other grade 2 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, conjunctival injection) on the ISO 11980 classification scale.
  14. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
  15. Any central corneal scar
  16. Any corneal distortion resulting from ocular diseases or previous hard or rigid gas permeable contact lens wear.
  17. Binocular vision abnormality, intermittent strabismus or strabismus.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai EENT Hospital, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 240 subjects were enrolled into this study. Of those enrolled, 199 subjects were randomized and dispensed one of the four study lenses while 41 subjects failed too meet all eligibility criteria. Of those dispensed, 14 subjects discontinued and 185 subjects completed all required study visits.
Groups:
- Test 1: Subjects randomized to receive senofilcon A (Test 1) lens throughout the entire duration of the study
- Test 2: Subjects randomized to receive senofilcon A (Test 2) throughout the entire duration of the study
- Test 3: Subjects randomized to receive senofilcon A (Test 3) throughout the entire duration of the study
- Control: Subjects randomized to receive the senofilcon A (Control) Lens throughout the entire duration of the study
Period: Overall Study
Arm/Group | Test 1 | Test 2 | Test 3 | Control
Started | 50 | 48 | 50 | 51
Completed | 49 | 45 | 44 | 47
Not Completed | 1 | 3 | 6 | 4
Not completed — Subject No Longer Meets Eligibility Criteria | 1 | 0 | 0 | 0
Not completed — Lens Discomfort | 0 | 1 | 0 | 0
Not completed — Unsatisfactory Visual Response due to Test Article | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lens Handling Difficulties | 0 | 0 | 1 | 0
Not completed — Subject Decided to Not Wear Contact Lenses | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Test 1: Subjects randomized to receive senofilcon A (Test 1) throughout the entire duration of the study
- Total: Total of all reporting groups
Arm/Group | Test 1 | Test 2 | Test 3 | Control | Total
Number analyzed (Participants) | 50 | 48 | 50 | 51 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (1.38) | 10.2 (1.51) | 10.0 (1.58) | 9.9 (1.59) | 10.0 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 24 | 25 | 106
  Male | 22 | 19 | 26 | 26 | 93
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Asian | 26 | 25 | 27 | 24 | 102
  Black or African American | 0 | 1 | 2 | 2 | 5
  White | 22 | 20 | 19 | 25 | 86
  Other | 2 | 2 | 2 | 0 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 3 | 5 | 4 | 17
  China | 25 | 24 | 25 | 23 | 97
  United States | 20 | 21 | 20 | 24 | 85

OUTCOME MEASURES:

1. Primary Outcome: Axial Length
Description: Axial length (in the unit of mm) was measured by a commercially available device based on the interferometry technique.
Time Frame: 6-month follow-up
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation was recorded.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | Test 1 | Test 2 | Test 3 | Control
Number analyzed (Participants) | 47 | 46 | 44 | 47
Number analyzed (eyes) | 94 | 92 | 88 | 94
mm | 0.119 (0.1008) | 0.135 (0.1165) | 0.079 (0.1251) | 0.189 (0.1206)
Statistical Analysis 1: Comparison: Test 1 vs Control; It was calculated that 160 participants randomized in a 1:1:1:1 fashion among the four arms would have at least 90% power to detect a 0.08 mm difference in mean axial elongation at the 6-month follow-up. The power analysis was conducted controlling 2-sided type I error of 0.05; Test type: Superiority — Superiority is established if the adjusted upper confidence limit is below 0; Mixed Models Analysis; The Kenward and Roger method was used for the denominator degrees of freedom; Mean Difference = -0.063, 95% CI 2-sided [-0.106 to -0.020], Standard Error of Mean 0.0181 — Mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Test 2 vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Superiority is established if the adjusted upper confidence limit is below 0; Mixed Models Analysis; The Kenward and Roger method was used for the denominator degrees of freedom; Mean Difference = -0.056, 95% CI 2-sided [-0.100 to -0.013], Standard Error of Mean 0.0183 — Mean difference was calculated as Test - Control
Statistical Analysis 3: Comparison: Test 3 vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Superiority is established if the adjusted upper confidence limit is below 0; Mixed Models Analysis; The Kenward and Roger method was used for the denominator degrees of freedom; Mean Difference = -0.105, 95% CI 2-sided [-0.149 to -0.062], Standard Error of Mean 0.0184 — Mean difference was calculated as Test - Control

2. Primary Outcome: Spherical Equivalent of Cycloplegic Autorefraction (SECAR)
Description: SECAR (in the unit of D) was computed from the spherocylindrical refraction measured by a commercially available autorefractor.
Time Frame: 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: D
Units Other Than Participants: eye
Arm/Group | Test 1 | Test 2 | Test 3 | Control
Number analyzed (Participants) | 47 | 46 | 44 | 47
Number analyzed (eye) | 94 | 92 | 88 | 94
D | -0.26 (0.32) | -0.25 (0.35) | -0.12 (0.27) | -0.35 (0.33)
Statistical Analysis 1: Comparison: Test 1 vs Control; It was calculated that 160 participants randomized in a 1:1:1:1 fashion among the four arms would have at least 79% power to detect a 0.20 D difference in mean axial elongation at the 6-month follow-up. The power analysis was conducted controlling 2-sided type I error of 0.05; Test type: Superiority — Superiority is established if the adjusted lower confidence limit is above 0; Mixed Models Analysis; Kenward and Roger method was for the denominator degrees of freedom; Mean Difference = 0.08, 95% CI 2-sided [-0.04 to 0.21], Standard Error of Mean 0.053 — Mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Test 2 vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Superiority is established if the adjusted lower confidence limit is above 0; Mixed Models Analysis; Kenward and Roger method was used for the denominator degrees of freedom; Mean Difference = 0.12, 95% CI 2-sided [-0.01 to 0.25], Standard Error of Mean 0.054 — Mean difference was calculated as Test - Control
Statistical Analysis 3: Comparison: Test 3 vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Superiority is established if the adjusted lower confidence limit is above 0; Mixed Models Analysis; Kenward and Roger method was used for the denominator degrees of freedom; Mean Difference = 0.22, 95% CI 2-sided [0.09 to 0.35], Standard Error of Mean 0.054 — Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study, 6-month up to 1 year.
Arm/Group | Test 1 | Test 2 | Test 3 | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/48 | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/48 | 1/50 | 0/51
Other Adverse Events (participants affected / at risk) | 9/50 | 4/48 | 2/50 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1 (N=50) | Test 2 (N=48) | Test 3 (N=50) | Control (N=51)
Cellulitis of Left Elbow and Upper Arm (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Mycoplasma Acute Bronchitis , Leukopenia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1 (N=50) | Test 2 (N=48) | Test 3 (N=50) | Control (N=51)
Cold (General disorders) | 9 (10) | 4 (5) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03408444/Prot_SAP_000.pdf